CLINICAL TRIAL: NCT05143827
Title: Glycemic Index of Pasta From Traditional and Current Wheat Varieties in Patients With Type 2 Diabetes: a Randomized, Cross-over, Blind Study
Brief Title: Glycemic Index of Pasta From Traditional and Current Wheat Varieties
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Edoardo Mannucci, Director, Diabetology unit, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 15425-IGGA1
Record Dates: First submitted 2021-11-23; First posted 2021-12-03 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Senatore Cappelli pasta (Experimental)
  Interventions: Other: Pasta manufactured with traditional wheat varieties (Senatore Cappelli, Korasan)
- Korasan pasta (Experimental)
  Interventions: Other: Pasta manufactured with traditional wheat varieties (Senatore Cappelli, Korasan)
- Claudio pasta (Active Comparator)
  Interventions: Other: Pasta manufactured with current wheat varieties (Claudio)

INTERVENTIONS:
Other: Pasta manufactured with traditional wheat varieties (Senatore Cappelli, Korasan) — A single meal composed of a portion of pasta (with standardized dressing) manufactured with different wheat varieties
  Arms: Korasan pasta; Senatore Cappelli pasta
Other: Pasta manufactured with current wheat varieties (Claudio) — A single meal composed of a portion of pasta (with standardized dressing) manufactured with different wheat varieties
  Arms: Claudio pasta

SUMMARY:
This randomized, cross-over study compares pasta produced with three different wheat varieties (Senatore Cappelli, Korasan, Claudio). Patients with type 2 diabetes with no pharmacological treatment will be randomized to three different sequences, and asked to eat a standard portion of pasta on three different occasions, four days apart. 3-hour post-prandial interstitial glucose profiles will be recorded using trans-cutaneous sensors.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Body Mass Index (BMI) > 20 kg/m2
* HbA1c < 58 mmol/mol

Exclusion Criteria:

* Current pharmacological therapy for diabetes (of any kind)
* Pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-20 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
60-min glucose | 60 minutes
  Glucose (interstitial monitoring) 60 min after beginning of meal

SECONDARY OUTCOMES:
30-min glucose | 30 minutes
  Glucose (interstitial monitoring) 30 min after beginning of meal
90-min glucose | 90 minutes
  Glucose (interstitial monitoring) 90 min after beginning of meal
120-min glucose | 120 minutes
  Glucose (interstitial monitoring) 120 min after beginning of meal
150-min glucose | 150 minutes
  Glucose (interstitial monitoring) 150 min after beginning of meal
180-min glucose | 180 minutes
  Glucose (interstitial monitoring) 180 min after beginning of meal
Area Under the Curve (AUC) glucose 30 min | 30 minutes
  Area under glucose (interstitial monitoring) curve 30 min after beginning of meal
AUC glucose 60 min | 60 minutes
  Area under glucose (interstitial monitoring) curve 60 min after beginning of meal
AUC glucose 90 min | 90 minutes
  Area under glucose (interstitial monitoring) curve 90 min after beginning of meal
AUC glucose 120 min | 120 minutes
  Area under glucose (interstitial monitoring) curve 120 min after beginning of meal
AUC glucose 180 min | 180 minutes
  Area under glucose (interstitial monitoring) curve 180 min after beginning of meal

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetologia AOU Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No